CLINICAL TRIAL: NCT06016283
Title: The Impact of Donor and Recipient Sex on Long-term Outcomes Following Living Donor Kidney Transplantation
Brief Title: Sex Impact on Long-term Outcomes of LDKT
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Yitian Fang, MD, MD, Erasmus Medical Center
Other Study IDs: Sex impact on LDKT
Record Dates: First submitted 2023-08-22; First posted 2023-08-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant Failure and Rejection; Gender
Keywords: gender; kidney transplantation; minor histocompatibility; graft survival
MeSH Terms: conditions — Rejection, Psychology; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- MDMR: Male recipient receiving kidney graft from male donor
- FDMR: Male recipient receiving kidney graft from female donor
- MDFR: Female recipient receiving kidney graft from male donor
- FDFR: Female recipient receiving kidney graft from female donor

SUMMARY:
The impact of donor and recipient gender combination on kidney transplant outcomes has been reported in several studies. The results vary greatly due to different factors, such as minor histocompatibility antigens, nephron overload, sex hormones, etc. Despite advancements in clinical practice, no large-scale studies exploring this question in living donor kidney transplantation have been conducted in the subsequent two decades. Our study aims to address this research gap and provide updated information on outcomes in relation to the gender combination following living donor kidney transplantation.

DETAILED DESCRIPTION:
The impact of donor and recipient gender combination on kidney transplant outcomes has been reported in several studies, but with inconclusive results. From an immunologic perspective, the transplantation of male donor kidneys into female recipients was associated with an increased risk of graft failure and mortality due to H-Y minor histocompatibility antigens. Another theory, based on nephron overload and hyperfiltration, suggests that male recipients of female donor kidneys tend to experience worse outcomes due to the smaller size of female kidneys. Additionally, the influence of sex hormones has been explored. Aufhauser et al. found that estrogen acts as a protective factor against ischemia-reperfusion injury (IRI), resulting in a significantly lower incidence of delayed graft function (DGF) in female recipients compared to male recipients. These findings seem conflicting, and most of studies have primarily focused on deceased donor kidney transplantation.

In addition, Kayler et al. analyzed a transplant database encompassing 30,258 living donor kidney transplantations between 1990 and 1999. Their study revealed a significant advantage in graft survival for male recipients of male donor kidneys compared to the other combinations. Another study involving 5,716 HLA-identical sibling kidney transplantations between 1985 and 2000 demonstrated that female recipients tend to have better graft survival rates regardless of the donor's gender. Despite advancements in clinical practice, no such large-scale studies exploring this question have been conducted in the subsequent two decades. Our study aims to address this research gap and provide updated information on outcomes in relation to the gender combination following living donor kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing living donor kidney transplantation in the Erasmus Medical Center between January 2010 and December 2020.

Exclusion Criteria:

* Recipients who were under 18 years at transplant or had no follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on biological gender.
Study Population: Patients undergoing living donor kidney transplantation in the Erasmus Medical Center between January 2010 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 1276 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Death-censored graft survival | From the date of kidney transplantation until the date of graft loss from any cause or the end of follow-up, whichever came first, assessed up to 10 years.
  Graft failure is defined as return to dialysis, transplant nephrectomy or retransplant. Death-censored graft failure was defined as the time from transplant to graft failure, with censoring for death with a functioning graft.

SECONDARY OUTCOMES:
Patient survival | From the date of kidney transplantation until the date of death from any cause or the end of follow-up, whichever came first, assessed up to 10 years.
  All-cause mortality is included in the patient survival.
DGF | From the date of kidney transplantation till the end of first posttransplant week, assessed up to one week.
  Delayed graft function (DGF) is defined as either the need for dialysis or the failure of a fall in serum creatinine of 10% on three consecutive days in the first posttransplant week.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Minnee, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Yitian Fang, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
The data that support this study are not publicly available due to the reasons of sensitivity and are available from the corresponding author upon reasonable request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT06016283/Prot_SAP_000.pdf